CLINICAL TRIAL: NCT03668379
Title: An Adaptive Treatment Intervention for Depression and Engagement in HIV Care Among Latinos Living With HIV
Brief Title: An Adaptive Intervention for Depression Among Latinos Living With HIV
Acronym: Latino-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: K01MH113475 (NIH); K01MH113475 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-09-12 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Depression
Keywords: Depression; HIV; Latinos; Sequential multiple assignment randomized trial designs; Mobile health; Cognitive-behavioral therapy
MeSH Terms: conditions — Depression | interventions — Maintenance; Telemedicine

STUDY DESIGN:
Intervention Model Description: The study utilizes a Sequential Multiple Assignment Randomized Trial (SMART) design in order to guide a series of adaptive behavioral interventions. In a SMART, eligible participants will be randomized at baseline and assigned to "1st-stage treatments" consisting of either 1. Behavioral Activation Therapy (BAT) or 2. BAT & mHealth. During the first stage treatment, Patient Health Questionnaire-9 (PHQ-9) scores will be collected. At the follow-up period, the PHQ-9 will provide a cutoff score to determine whether a participant showed a clinically meaningful response ("responder/non-responder") to the "1st stage treatment." "Responder" indicates that patients successfully responded to the 1st stage treatment and will continue the treatment in maintenance mode. "Non-responder" indicates that the patient did not respond to the 1st-stage treatment and are re-randomized to either an augmented or "switched" intervention.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Medical providers of the patients enrolled in the study will be notified that their patient is in a study for depression but not told what intervention arm. At all follow-up outcome points, the assessor will be blind to all intervention arms the patient were randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation Therapy (Active Comparator): During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of five, 1-hour sessions will be delivered every two weeks. During Session 1, the focus will be on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 will review the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 will review progress, challenges & maintenance strategies.
  Interventions: Behavioral: Augment w/mHealth; Behavioral: Maintenance; Behavioral: Switch to CBT & mHealth
- Behavioral Activation Therapy & mHealth (Experimental): During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  Interventions: Behavioral: Maintenance; Behavioral: Switch to CBT & mHealth; Behavioral: Augment w/BAT & mHealth

INTERVENTIONS:
Behavioral: Augment w/mHealth — "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Arms: Behavioral Activation Therapy
Behavioral: Maintenance — "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
Behavioral: Switch to CBT & mHealth — "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
Behavioral: Augment w/BAT & mHealth — "Non-responders" to the BAT & mHealth intervention may be re-randomized to receive an additional "dose" of BAT & mHealth in the form of an additional session of BAT.
  Arms: Behavioral Activation Therapy & mHealth

SUMMARY:
This study will use a pilot sequential multiple assignment randomized trial (SMART) design to build an adaptive treatment strategy (ATS) for depression and engagement in HIV among Latinos living with HIV. The ATS is the sequencing of treatments, which are a behavioral activation therapy (BAT), a cognitive-behavioral therapy (CBT), and mobile health (mHealth) tool. The outcomes are to assess the feasibility of the SMART and ATS in the HIV care site and acceptability of the SMART and ATS to patients and clinic staff.

DETAILED DESCRIPTION:
This project proposes to use a SMART to build an adaptive treatment strategy (ATS) that has a mobile health (mHealth) tool (text-messaging) to improve adherence to the treatments for depression. The treatments being tested are a behavioral activation therapy (BAT) and cognitive-behavioral therapy (CBT). The outcomes are feasibility of the SMART and ATS in the HIV care site and acceptability of the SMART and ATS to patients and clinic staff. To achieve the overall goal, there are two aims. Aim 1 uses qualitative research methods for the conduct of focus groups and individual interviews with HIV+ Latinos in both English and Spanish. The goal of Aim 1 is to tailor the intervention to the cultural and linguistic needs of Latinos and the organization needs of the HIV clinic study site, which informs Aim 2. Aim 1 is guided by the CDCs Map of Adaptation tailoring framework, which consist of three Action Steps. Action Step 1-3 are to better understand and document: 1) expressions for depression in Spanish and barriers to care, 2) language issues in detecting and reporting depressive symptoms, 3) cultural perspectives of how depression presents as a barrier to care, and 4) attitudes (i.e., cognitive and emotional evaluations) toward BAT and CBT, and text-message preference and confidentiality concerns to promote adherence to the intervention activities. Aim 2 is to build and test a pilot SMART for an ATS - a set of decision rules that uses detectable changes in patient health status to inform the next course of treatment. Successful completion of the proposed study will yield pilot data on the feasibility and acceptability of an ATS for depression integrated into HIV primary care at the University of California San Francisco - Zuckerberg San Francisco General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* 18 years of age and older
* Self identifies as Latino/Hispanic
* Fluent in English or Spanish
* Receives HIV care at study site clinic
* Has a moderate depression severity score or higher (Patient Health Questionnaire-9 score >9; PHQ)
* Agrees to discuss depression, treatment preferences, and mobile health
* Owns a mobile phone that can send/receive short-message service (SMS) text messages
* Agrees to participate in the intervention that lasts three months
* Agrees to have medical and clinical data abstracted one year after baseline
* Able and willing to consent to participate

Exclusion Criteria:

* Not HIV positive
* Under 18 years of age
* Does not self-identify as Latino/Hispanic
* Not fluent in English or Spanish
* Does not receive primary HIV care at the study site
* Has a less than moderate depression severity score (Patient Health Questionnaire-9 score ≤9; PHQ)
* Does not agree to discuss depression, treatment preferences, and mobile health
* Does not owns a mobile phone that can send/receive short-message service (SMS) text messages
* Does not agree to participate in the intervention that lasts three months
* Does not agree to have medical and clinical data abstracted one year after baseline
* Not able and willing to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Sauceda, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ward 86 HIV Clinic, Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfeiffer PN, Bohnert KM, Zivin K, Yosef M, Valenstein M, Aikens JE, Piette JD. Mobile health monitoring to characterize depression symptom trajectories in primary care. J Affect Disord. 2015 Mar 15;174:281-6. doi: 10.1016/j.jad.2014.11.040. Epub 2014 Nov 28. PMID 25527999
- [Background] Almirall D, Compton SN, Gunlicks-Stoessel M, Duan N, Murphy SA. Designing a pilot sequential multiple assignment randomized trial for developing an adaptive treatment strategy. Stat Med. 2012 Jul 30;31(17):1887-902. doi: 10.1002/sim.4512. Epub 2012 Mar 22. PMID 22438190
- [Background] Hopko DR, Lejuez CW, Ruggiero KJ, Eifert GH. Contemporary behavioral activation treatments for depression: procedures, principles, and progress. Clin Psychol Rev. 2003 Oct;23(5):699-717. doi: 10.1016/s0272-7358(03)00070-9. PMID 12971906
- [Background] Safren SA, O'Cleirigh C, Tan JY, Raminani SR, Reilly LC, Otto MW, Mayer KH. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in HIV-infected individuals. Health Psychol. 2009 Jan;28(1):1-10. doi: 10.1037/a0012715. PMID 19210012
- [Background] Christopoulos KA, Riley ED, Tulsky J, Carrico AW, Moskowitz JT, Wilson L, Coffin LS, Falahati V, Akerley J, Hilton JF. A text messaging intervention to improve retention in care and virologic suppression in a U.S. urban safety-net HIV clinic: study protocol for the Connect4Care (C4C) randomized controlled trial. BMC Infect Dis. 2014 Dec 31;14:718. doi: 10.1186/s12879-014-0718-6. PMID 25551175
- [Background] Murphy SA, Lynch KG, Oslin D, McKay JR, TenHave T. Developing adaptive treatment strategies in substance abuse research. Drug Alcohol Depend. 2007 May;88 Suppl 2(Suppl 2):S24-30. doi: 10.1016/j.drugalcdep.2006.09.008. Epub 2006 Oct 23. PMID 17056207
- [Background] Dimidjian S, Barrera M Jr, Martell C, Munoz RF, Lewinsohn PM. The origins and current status of behavioral activation treatments for depression. Annu Rev Clin Psychol. 2011;7:1-38. doi: 10.1146/annurev-clinpsy-032210-104535. PMID 21275642
- [Background] Simoni JM, Wiebe JS, Sauceda JA, Huh D, Sanchez G, Longoria V, Andres Bedoya C, Safren SA. A preliminary RCT of CBT-AD for adherence and depression among HIV-positive Latinos on the U.S.-Mexico border: the Nuevo Dia study. AIDS Behav. 2013 Oct;17(8):2816-29. doi: 10.1007/s10461-013-0538-5. PMID 23812892
- [Background] McKleroy VS, Galbraith JS, Cummings B, Jones P, Harshbarger C, Collins C, Gelaude D, Carey JW; ADAPT Team. Adapting evidence-based behavioral interventions for new settings and target populations. AIDS Educ Prev. 2006 Aug;18(4 Suppl A):59-73. doi: 10.1521/aeap.2006.18.supp.59. PMID 16987089

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation Therapy: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of five, 1-hour sessions will be delivered every two weeks. During Session 1, the focus will be on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 will review the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 will review progress, challenges & maintenance strategies.
  If participants responded to the intervention, they will continue with stage 1 treatment. This means that they will stay the course with the current assignment, which means finishing three more sessions, which makes the overall total of eight sessions.
- Behavioral Activation Therapy & mHealth: During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  If participants responded to the intervention, they will continue with stage 1 treatment. This means that they will stay the course with the current assignment, which means finishing three more sessions, which makes the overall total of eight sessions.
- Behavioral Activation Therapy Augment With mHealth: This arm included participants who did not respond to BAT in stage 1.
  In stage 1, a trained graduate student provided five weekly BAT sessions. Session 1, the focus was on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 reviewed the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 reviewed progress, challenges & maintenance strategies.
  "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention in the second stage.
- Behavioral Activation Therapy Switch to Cognitive Behavioral Therapy & mHealth: This arm included participants who did not respond to BAT in stage 1.
  In stage 1, a trained graduate student provided five weekly BAT sessions. Session 1, the focus was on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 reviewed the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 reviewed progress, challenges & maintenance strategies.
  "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
- Behavioral Activation Therapy & mHealth Switch to Cognitive Behavioral Therapy & mHealth: This arm included participants who did not respond to BAT & mHealth.
  In stage 1, a trained graduate student provided five weekly BAT sessions.
  During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
- Behavioral Activation Therapy & mHealth Augment With Behavioral Activation Therapy & mHealth: This arm included participants who did not respond to BAT and BAT & mHealth.
  In stage 1, a trained graduate student provided five weekly BAT sessions.
  During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  "Non-responders" to the BAT & mHealth intervention may be re-randomized to receive an additional "dose" of BAT & mHealth in the form of an additional session of BAT.
Period: Stage 1 Intervention (Months 1-2)
Arm/Group | Behavioral Activation Therapy | Behavioral Activation Therapy & mHealth | Behavioral Activation Therapy Augment With mHealth | Behavioral Activation Therapy Switch to Cognitive Behavioral Therapy & mHealth | Behavioral Activation Therapy & mHealth Switch to Cognitive Behavioral Therapy & mHealth | Behavioral Activation Therapy & mHealth Augment With Behavioral Activation Therapy & mHealth
Started | 5 | 5 | 0 | 0 | 0 | 0
Completed | 4 | 3 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0
Period: Stage 2 Intervention (Months 3-4)
Arm/Group | Behavioral Activation Therapy | Behavioral Activation Therapy & mHealth | Behavioral Activation Therapy Augment With mHealth | Behavioral Activation Therapy Switch to Cognitive Behavioral Therapy & mHealth | Behavioral Activation Therapy & mHealth Switch to Cognitive Behavioral Therapy & mHealth | Behavioral Activation Therapy & mHealth Augment With Behavioral Activation Therapy & mHealth
Started | 4 | 3 | 0 | 0 | 0 | 0
Completed | 3 | 1 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Activation Therapy: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of eight, 1-hour sessions will be delivered every two weeks.
  Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation Therapy | Behavioral Activation Therapy & mHealth | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (12.5) | 48.4 (14.5) | 47 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 is a self-report measure of depression with a range from 0-27, with higher score indicating greater severity of depression symptoms.
  units on a scale | 10.2 (3.7) | 13.6 (4.21) | 11.9 (4.14)
The Index of HIV Care Engagement-- or index of [Mean (Standard Deviation); unit: units on a scale] — This Index measures perceived engagement and connection to HIV care. Scores are the sum of all 10 items with response options being 1 to 5. Sum scores are then divided by 10 with a range of 1-5. The higher scores indicate better engagement in care.
  units on a scale | 4.24 (0.84) | 4.15 (0.60) | 4.20 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Composite Measure of Feasibility for the Adaptive Treatment Strategy (ATS)
Description: This is one composite measure. Feasibility of the adaptive treatment strategy (ATS) will be measured to assess whether the ATS is appropriate for further testing, relevant and sustainable. Feasibility of the ATS will be reported as a composite score of the following measures taken at the end of the second-stage treatment:
  1. Total number of participants screened, eligible and enrolled;
  2. At least 80% of all BAT & CBT sessions completed;
  3. 80% retention of participants across all "outcome groups".
Time Frame: 4 months
Population: In this study, all participants assigned to their 1st stage treatment either responded and entered the maintenance arm or did not complete the intervention. Thus, we had no non-responders and no re-randomized participants who would have either augmented or changed their 1st stage treatment. Results reflect this result and zero cells in the other arms.
Measure: Count of Participants; unit: Participants
Groups:
- Behavioral Activation Therapy Maintenance: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of eight, 1-hour sessions will be delivered every two weeks. D Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
- Behavioral Activation Therapy & mHealth Maintenance: During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
  Augment w/BAT & mHealth: "Non-responders" to the BAT & mHealth intervention may be re-randomized to receive an additional "dose" of BAT & mHealth in the form of an additional session of BAT.
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 5 | 5
Participants
  Enrolled | 5 | 5
  Completion Percentage | 4 | 3
  Retention Percentage | 0 | 0

2. Primary Outcome: Composite Measure of Acceptability for the Adaptive Treatment Strategy (ATS)
Description: This is one composite measure. Acceptability of the adaptive treatment strategy will be measured to determine the tolerability or appropriateness of the SMART intervention from the perspective of both participants and clinicians.Acceptability of the ATS will be reported as a composite score of the following measures taken at the end of the second-stage treatment:
  1. Greater than 90% adherence to the BAT & CBT session schedule;
  2. Responsiveness to text-messages: a) >80% of all two-way messages replied back to study line during the set of blocked hours; b) >90% of participants reporting direct benefit from one-way text messages;
  3. Acceptability responses coded from post-intervention exit interview transcripts;
  4. Limited number of barriers to participation reported by participants in exit interviews;
  5. Responses to a brief survey (to be developed) assessing clinic staff acceptability of the intervention.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Behavioral Activation Therapy Maintenance: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of eight, 1-hour sessions will be delivered every two weeks.
  Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 5 | 5
Participants
  90% Adherence | 3 | 1
  Two-Way Text-Message Response | 0 | 0
  One-Way Text-Message Response | 0 | 0
  Acceptability Responses | 0 | 0
  Barriers | 0 | 0
  Responses | 0 | 0

3. Secondary Outcome: Self-reported Adherence to Antiretroviral Therapy (ART)
Description: Self-reported adherence will be measured using the the visual analog scale (VAS), a 10-cm line on which participants indicate the percentage of doses (intervals of 10 percentage points indicated from 0% to 100%) of all HIV medications taken in the past 30 days (Amico et al., 2006). Higher percentage indicates greater adherence to HIV medications. This measure will be used for descriptive purposes.
Time Frame: 12 months
Population: The disruptions of COVID-19 prevented us from collecting data 12-month survey data and thus, we have entered "0" into the cells as instructed.
Groups:
- Behavioral Activation Therapy Maintenance: The initial stage treatment is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of five, 1-hour sessions will be delivered every two weeks. During Session 1, the focus will be on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 will review the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 will review progress, challenges & maintenance strategies.
  Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Viral Load
Description: Viral load measures the amount of HIV virus in the blood. Viral load data abstracted from patient medical records will act as a descriptive measure of HIV-related clinical outcomes. A detectable viral load is a measurement of the amount of HIV in the blood, and an indication that HIV is replicating in the body. Undetectable viral load means that there is not enough of the virus to be detected.
Time Frame: 12 months
Population: We could not abstract viral load data from 1 participant.
Measure: Number; unit: participants
Groups:
- Behavioral Activation Therapy Maintenance: The initial stage treatment, is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of five, 1-hour sessions will be delivered every two weeks. During Session 1, the focus will be on providing an introduction to BAT, as well as building "confianza" (mutual trust) between the patient and provider. Sessions 2 & 3 will review the initial session, introduce "high" value activities and barriers to BAT protocols. Sessions 4 & 5 will review progress, challenges & maintenance strategies.
  Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 4 | 5
participants
  Undetectable viral load | 3 | 4
  Detectable viral load | 1 | 1

5. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Patient Health Questionnaire-9 is a self-report measure of depression with a range from 0-27, with higher score indicating greater severity of depression symptoms.
Time Frame: 12 months
Population: as for outcome 3
Groups:
- Behavioral Activation Therapy Maintenance: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program intervention. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of eight, 1-hour sessions will be delivered every two weeks. D Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
- Behavioral Activation Therapy & mHealth Maintenance: During the initial stage treatment, the experimental arm will deliver a BAT program identical to the active comparator arm, as well as a mobile health (mHealth) component in the form of one-way and two-way SMS text-messages. Direct personalized text-messages will be delivered twice a week to facilitate engagement with the BAT intervention activities. One-way messages will be sent as appointment and BAT adherence reminders. Two-way messages will be sent once a week during a set block of protected hours, creating a "mobile drop-in clinic" where messages can be sent and received.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Engagement in HIV Care
Description: Engagement in care will be measured utilizing the multidimensional index of engagement in HIV care, a 10-item unit-dimensional patient-centered scale that assesses provider, clinic, and patient-level characteristics associated with being engaged in HIV care. This measure will be used for descriptive purposes. Mean scores are the sum of all 10 items divided by 10 with a range of 1-5, and higher scores indicate better engagement in care.
Time Frame: 12 months
Population: as for outcome 3
Arm/Group | Behavioral Activation Therapy Maintenance | Behavioral Activation Therapy & mHealth Maintenance
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Description: An adverse event is any unfavorable or unintended disease, sign, or symptom that is temporally associated with the use of the intervention. An adverse event may or may not be considered related to the intervention or study procedures. Such events can be related to the intervention, dose, or route of administration.
Groups:
- Behavioral Activation Therapy: During the initial stage treatment, the active comparator arm is the behavioral activation (BAT) program. BAT is informed by behavioral theory and has been shown to be a highly efficacious treatment for depression. A total of eight, 1-hour sessions will be delivered every two weeks.
  Augment w/mHealth: "Non-responders" to the first stage treatment of BAT alone may be re-randomized to this augmented intervention to receive text-message support in addition to the BAT intervention.
  Maintenance: "Responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth will continue in maintenance mode. These participants will not receive any additional interventions during the 2nd-stage treatment.
  Switch to CBT & mHealth: "Non-responders" to the 1st-stage treatment of either 1. BAT or 2. BAT & mHealth may be re-randomized to "switch" interventions in the form of an intensified "dose" of Cognitive Behavioral Therapy (CBT). CBT is eight sessions long and covers five modules that can be re-arranged to fit patient needs. Sessions will be scheduled once a week to facilitate more contact with participants. An identical text-messaged tool will be used.
Arm/Group | Behavioral Activation Therapy | Behavioral Activation Therapy & mHealth
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The trial was severely limited by COVID-19. The trial launched recruitment in late February 2020, and the University of California, San Francisco instituted a complete pausing of non-essential research in March of 2020. This was followed by ongoing pauses and delays with each new COVID-19 variants and corresponding restrictions, such as limited capacity of to engage with participants given social distancing policies on site. Each part of the trial was severely limited and negatively impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03668379/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03668379/ICF_001.pdf